CLINICAL TRIAL: NCT01245101
Title: A Prospective, Open-Label, Double-Arm, Crossover, Single-Center Pilot Study to Evaluate the Addition of Raltegravir to Established Suppressive Antiretroviral Therapy While Monitoring Changes in Markers of Immune Activation Among HIV-1 Infected Individuals Without Adequate Immune Restoration
Brief Title: Addition of Raltegravir to Established Antiretroviral Suppressive Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: University of Miami (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Rafael Campo, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20100499
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: HIV
Keywords: HIV raltegravir intensification replication activation
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir and then Observation (Experimental): The total duration of the study will be 40 weeks. This will include Part 1 (16 weeks) followed by Part 2 (8 weeks) followed by the crossover to Part 2 (16 weeks). During Part 1 participants in Group A will receive open-label raltegravir in addition to their established antiretroviral regimen while Group B participants will continue taking their established antiretroviral regimen for 16 weeks. After completion of Part 1, both groups will enter Part 2 that will consist of a washout period of 8 weeks during which both groups will only take their established antiretroviral regimen without raltegravir. This will be followed by Part 3 during which the two study groups will undergo a crossover with respect to the treatment assignment during Part 1 so that Group A will continue to receive their established antiretroviral regimen while Group B will receive open-label raltegravir in addition to their established antiretroviral regimen for 16 weeks.
  Interventions: Drug: Raltegravir
- Observation and then Raltegravir (Active Comparator): The total duration of the study will be 40 weeks. This will include Part 1 (16 weeks) followed by Part 2 (8 weeks) followed by the crossover to Part 2 (16 weeks). During Part 1 participants in Group A will receive open-label raltegravir in addition to their established antiretroviral regimen while Group B participants will continue taking their established antiretroviral regimen for 16 weeks. After completion of Part 1, both groups will enter Part 2 that will consist of a washout period of 8 weeks during which both groups will only take their established antiretroviral regimen without raltegravir. This will be followed by Part 3 during which the two study groups will undergo a crossover with respect to the treatment assignment during Part 1 so that Group A will continue to receive their established antiretroviral regimen while Group B will receive open-label raltegravir in addition to their established antiretroviral regimen for 16 weeks.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg twice daily in addition to subject's antiretroviral therapy.
  Arms: Raltegravir and then Observation
Drug: Raltegravir — Raltegravir 400 mg twice daily in addition to subject's antiretroviral therapy.
  Arms: Observation and then Raltegravir

SUMMARY:
This study will examine whether intensification with raltegravir of a suppressive antiretroviral regimen in HIV infected patients with poor immune restoration has a beneficial effect on cryptic viral replication and the immune system. Specifically, the investigators will examine the effect that raltegravir intensification of ART has on episomal cDNA frequencies, immune activation, CD4+ cell counts and apoptosis, and markers of microbial translocation.

DETAILED DESCRIPTION:
This is a single-center, open-label, double-arm, crossover study which will include approximately 40 HIV-infected subjects on an established suppressive HAART for at least 2 years with evidence of undetectable HIV-1 RNA levels (either <50 copies/ml by RT-PCR or <75 copies/ml by bDNA assay) and CD4+ count of <350 cells/mm3 or an increase in CD4+count <100 cells/mm3 in the last 2 years. Participants (~20 Group 1 and ~20 in Group 2) will be randomly assigned to 1 of the 2 treatment arms described below in Table 1:

Table 1. Study groups and treatment assignments

Group A Raltegravir 400 mg PO q12h in addition to established ART (Part 1) followed by a washout period only on ART (Part 2) followed by ART (Part 3)

Group B Established ART (Part 1) followed by a washout period only on ART (Part 2) followed by raltegravir 400 mg PO q12h in addition to ART (Part 3)

The participants' pre-study HAART will be monitored so as to ensure that the distribution of NNRTI to PI-based regimens is roughly 1:1 and no higher than 2 (NNRTI):1 (PI).

The total duration of the study will be 40 weeks. This will include Part 1 (16 weeks) followed by Part 2 (8 weeks) followed by the crossover to Part 2 (16 weeks) (Figure 1). During Part 1 participants in Group A will receive open-label raltegravir in addition to their established antiretroviral regimen while Group B participants will continue taking their established antiretroviral regimen for 16 weeks. After completion of Part 1, both groups will enter Part 2 that will consist of a washout period of 8 weeks during which both groups will only take their established antiretroviral regimen without raltegravir. This will be followed by Part 3 during which the two study groups will undergo a crossover with respect to the treatment assignment during Part 1 so that Group A will continue to receive their established antiretroviral regimen while Group B will receive open-label raltegravir in addition to their established antiretroviral regimen for 16 weeks.

After obtaining informed consent, patients will be enrolled into the study, a study number will be assigned, a complete history will be obtained, and a physical exam will be performed. Blood will be drawn for the following laboratory exams at Day 1 and at Weeks 1, 2, 4, 10, 16, 24, 25 26, and 40 for Group A and at Day 1 and at Weeks 1, 2, 16, 24, 25, 26, 28, 34, and 40 for Group B:

* T-cell subsets
* Plasma viral load
* Episomal viral cDNA PCR
* HLA-DR levels
* CD38 levels

Blood will also be drawn for the following laboratory exams at Day 1 and at Weeks 4, 12, 16, 24, 28, 36, and 40 for both Group A and Group B to determine

* Plasma levels of LPS, 16s ribosomal DNA, and sCD14
* T cell receptor excision circles
* CD4+ and CD8+ T-cell apoptosis

At all visits, a directed physical exam will be performed on an as-needed-basis.

ELIGIBILITY:
Inclusion Criteria:

To qualify for this study, participants will need to have:

1. At least 18 years of age
2. Documented HIV-1 infection
3. CD4+ count <350 cells/mm3 at the time of enrollment or CD4+ count increase of <100 cells/mm3 within the past 2 years
4. Plasma viral load <400 copies/ml at all testing time points within the preceding 2 years AND <50 copies/ml by RT-PCR or <75 copies/ml by bDNA at the 2 testing time points immediately preceding enrollment into the study

Exclusion Criteria:

To qualify for this study, patients must not meet any of the following exclusion criteria:

1. Pregnancy or breast-feeding
2. Prior use of raltegravir at any time in the past
3. Use of any investigational, immunomodulatory, immunosuppressive agents within 90 days prior or during this study
4. Alcohol or substance abuse that in the opinion of the investigator might interfere with patient compliance or safety
5. Any condition or pre-study laboratory abnormality that in the opinion of the investigator might interfere with patient compliance or safety

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael E Campo, MD, Principal Investigator — University of Miami
Locations (1):
- Infectious Diseases Research Unit, University of Miami Miller School of Medicine, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note: because of poor enrollment and inability to find the originally planned 40 patients, the study was terminated after only 15 of 20 planned patients had been enrolled into the Raltegravir Then Observation arm. No patients were enrolled into the Observation Then Raltegravir arm.
Groups:
- Raltegravir Then Observation: Raltegravir 400 mg twice a day for 16 weeks followed by a washout of 8 weeks followed by Observation of 16 weeks.
- Observation Then Raltegravir: Observation for 16 weeks followed by a washout of 8 weeks followed by Raltegravir 400mg twice a day for 16 weeks.
Period: Period 1 (Treatment)
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir
Started | 15 | 0
Completed | 13 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Period 2 (Washout)
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir
Started | 13 | 0
Completed | 12 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 3 (Treatment)
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir
Started | 12 | 0
Completed | 11 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir | Total
Number analyzed (Participants) | 15 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 13 |  | 13
  >=65 years | 2 |  | 2
Gender [Count of Participants; unit: Participants]
  Female | 11 |  | 11
  Male | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Episomal HIV cDNA Formation
Description: These are linear viral cDNAs that are subsequently circularized by the DNA repair apparatus of the host cell to form episomes. They are markers of ongoing viral replication.
Time Frame: 16 weeks
Population: 11 of 12 subjects meeting the per protocol definition were analyzed for the Raltegravir then Observation arm. Poor enrollment led to early termination of study before second arm was activated.
Measure: Mean (Standard Deviation); unit: copies/million
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir
Number analyzed (Participants) | 11 | 0
copies/million
  Raltegravir | 4.581 (13.72) |
  Observation | 0.7173 (1.02) |

2. Secondary Outcome: Markers of Immune Activation
Description: Flow cytometry will be performed in whole blood for analysis of markers of immune activation by standard methodology using a LSR-II flow cytometer. Percentage and absolute counts of CD8+CD38+ cells will be determined as the main outcome measure.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of activated CD8+CD38+ cells
Arm/Group | Raltegravir Then Observation | Observation Then Raltegravir
Number analyzed (Participants) | 11 | 0
Percentage of activated CD8+CD38+ cells
  Raltegravir | 22.37 (16.73) |
  Observation | 26.72 (14.93) |

ADVERSE EVENTS:
Groups:
- Raltegravir: Raltegravir 400 mg twice a day for 16 weeks
- Observation: Observation for 16 weeks
Arm/Group | Raltegravir | Observation
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/0
Other Adverse Events (participants affected / at risk) | 1/15 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=15) | Observation (N=0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only 11 of 12 patients completed week 40 and were analyzed as per protocol. In view of poor enrollment and a simple analysis of the limited amount of data that failed to support our hypothesis, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes